CLINICAL TRIAL: NCT03672240
Title: A Phase Ib Study of APL-1202 in NMIBC Patients Who Are Resistant to One Induction Course of BCG Treatment
Brief Title: Study of APL-1202 in Non-Muscle Invasive Bladder Cancer Patients Who Are Resistant to One Induction Course of BCG Treatment
Acronym: NMIBC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asieris Pharmaceutical Technologies Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: AsierisPharma (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YHGT-NB-01
Record Dates: First submitted 2018-09-05; First posted 2018-09-14 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Non-Muscle Invasive Bladder Cancer (NMIBC)
Keywords: Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Cancer (NMIBC); Oral Antineoplastic Agent
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APL-1202 (Experimental): * APL-1202 will be administered orally at daily 750 mg (250 mg, TID) for 5-7 days prior to the first intravesical BCG treatment and continue for additional 11 weeks (a total 12 weeks of dosing with APL-1202).
  * Standard intravesical BCG induction course (once weekly for 6 weeks) 50 mg TICE BCG in 50 mL sterile saline (or a full dose standard vial of BCG) will be initiated on Week 2.
  Interventions: Drug: APL-1202

INTERVENTIONS:
Drug: APL-1202 — To assess the safety and pharmacokinetics of APL-1202 alone and in combination with Bacillus Calmette Guerin

SUMMARY:
A Phase Ib, open label, non randomized study to measure the safety and PK characteristics of APL-1202 at steady-state in adult male and female BCG resistant NMIBC patients when it is administered alone and concurrently with BCG.

DETAILED DESCRIPTION:
Six eligible participants will be administered with APL-1202 one week prior to the first BCG instillation, during the six-week course of BCG instillation, and additional five weeks, for a total of 12 weeks of dosing. Safety assessment will be performed during the entire 13 week study duration. Plasma and urine samples will be collected from each participant at prior to first and fifth BCG instillations for PK analysis.

ELIGIBILITY:
Subject Eligibility Criteria:

Inclusion Criteria:

1. History of Intermediate Risk or High Risk Transitional Cell Carcinoma Non-Muscle Invasive Bladder Cancer as defined by AUA Guidelines:

   AUA Risk Stratification for Non-Muscle Invasive Bladder Cancer

   Low Risk LGa solitary Ta ≤ 3cm PUNLMPb

   Intermediate Risk Recurrence within 1 year Solitary LG Ta > 3cm LG Ta, multifocal HGc Ta, ≤ 3cm LG T1

   High Risk HG T1 Any recurrent, HG Ta HG Ta, >3cm (or multifocal) Any CISd Any BCG failure in HG patient Any variant histology Any LVIe Any HG prostatic urethral

   a. LG = low grade; b. PUNLMP = papillary urothelial neoplasm of low malignant potential; c. HG = high grade; d. CIS=carcinoma in situ; e. LVI = lymphovascular invasion.
2. History of prior induction course of intravesical BCG, using 1/3 to full dose of BCG for 6 treatments (BCG Naïve will not be eligible). Previous BCG treatment in combination with interferon is allowed.
3. Patients who are eligible will either receive maintenance course (3 treatments 1/3 to full dose) or repeat induction course (6 treatments 1/3 to full dose)
4. Principal Investigator's discretion if patients who have a negative cystoscopy or urine cytology following initial BCG induction, can be placed on maintenance BCG to recurrence of bladder cancer
5. 18 years of age or older
6. Eastern Cooperative Oncology Group (ECOG) performance status < 2
7. Not pregnant or lactating
8. Subjects with child bearing or fathering potential must agree to use adequate contraception during the study and for 3 months after last treatment of investigational drug
9. Agree to study specific informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information
10. Adequate baseline complete blood count (CBC), renal and hepatic function:

1) Parameters described as WBC > 3000 cells/mm3, ANC > 1,000 cells/mm3, hemoglobin > 8.5 g/dL, and platelet count >100,000 cells/mm3 2) Adequate renal function: serum creatinine < 1.5 x upper limit of normal (ULN) 3) Bilirubin, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) are not more than 2 x Upper Limits of Normal 4) Absolute lymphocyte count ≥ 800/μL before the first dose of APL-1202

Exclusion Criteria:

1. Stage T2 or above urothelial carcinoma or urothelial carcinoma outside the bladder
2. Stage T1 NMIBC recurred at 3 months or shorter from the first dose of prior induction BCG course
3. Recurrent high-grade Ta/T1 disease within 6 months from the last dose of adequate BCG therapy
4. Previous systemic immunotherapy for bladder cancer
5. Prior major surgery (not Transurethral Resection of Bladder Tumor [TURBT/Cystoscopy]), radiation therapy, or systemic therapy within 8 weeks of starting the study treatment
6. National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) Grade 3 hemorrhage within four weeks from the starting study treatment
7. Any of the following medical conditions within the six months prior to investigational drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
8. Hypertension that cannot be controlled by medications
9. Optic nerve disorders or with a history of optic nerve disorders
10. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or investigational drug administration, or may interfere with the interpretation of study results in the judgment of the Investigator
11. Clinically meaningful allergic reactions or any known hypersensitivity or prior reaction to any of the formulation components in the investigational drug
12. Systemic treatment on any investigational clinical trial within 28 days (or 5 half-lives of that agent, whichever is greater) prior to enrollment
13. Concurrent treatment with immunosuppressive or immunomodulatory agents, including any systemic steroid (exception: inhaled or topically applied steroids, and acute and chronic standard dose nonsteroidal anti-inflammatory drugs (NSAIDs), are permitted). Use of a short course (i.e., ≤ 2 day) of a glucocorticoid is acceptable to prevent a reaction to the IV contrast used for: computed tomography (CT) scans
14. Immunosuppressive therapy, including: cyclosporine, anti-thymocyte globulin, or tacrolimus within three months of study entry
15. Concurrent treatment with strong inducers or inhibitors of CYP450 enzymes
16. Concurrent treatment with low therapeutic index drugs (such as methotrexate) that are renally cleared by OAT1- and OAT3-mediated transport
17. History of prior malignancy, except for adequately treated in situ cancer or basal cell or squamous cell skin cancer or other cancers (e.g. breast, prostate) for which the patient has been disease free and/or received curative therapy. Exclusion of patients described above will be at the discretion of the Sponsor.
18. Progressive or persistent viral or bacterial infection
19. All infections must be resolved, and the subject must remain afebrile for seven days without antibiotics prior to enrollment
20. Urinary tract infection, including particularly bladder infection, must be resolved prior to being placed on study
21. Unmanageable active gastric ulcer or inflammation of gastrointestinal (GI) tract
22. Gastric bleeding within last 6 months prior to enrollment
23. Anuria
24. Unable to take oral medication
25. Unwilling or unable to comply with the protocol or cooperate fully with the Investigator and site personnel
26. Unwilling to sign the informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Treatment-Related Adverse Events | 13 weeks
  Incidence and Severity of Treatment-Related Adverse Events as Assessed by CTCAE v.5.0 or newer

SECONDARY OUTCOMES:
Pharmacokinetics - Area Under Curve | On Week 2 prior to first BCG instillation
  PK measurement expressed as area under curve for APL-1202
Pharmacokinetics - Area Under Curve | On Week 6 prior to fifth BCG instillation
  PK measurement expressed as area under curve for APL-1202
Pharmacokinetics - Maximum Plasma Concentration | On Week 2 prior to first BCG instillation
  PK measurement expressed as maximum plasma concentration for APL-1202
Pharmacokinetics - Maximum Plasma Concentration | On Week 6 prior to fifth BCG instillation
  PK measurement expressed as maximum plasma concentration for APL-1202
Pharmacokinetics - Half-Life | On Week 2 prior to first BCG instillation
  PK measurement expressed as half-life for APL-1202
Pharmacokinetics - Half-Life | On Week 6 prior to fifth BCG instillation
  PK measurement expressed as half-life for APL-1202
Pharmacokinetics - Cumulative Amount in Urinary Excretion | Eight hours after first dose on Week 2 prior to first BCG instillation
  PK measurement expressed as cumulative amount in urinary excretion for APL-1202
Pharmacokinetics - Cumulative Amount in Urinary Excretion | Eight hours after first dose on Week 6 prior to fifth BCG instillation
  PK measurement expressed as cumulative amount in urinary excretion for APL-1202
Pharmacokinetics - Cumulative Fraction of Dose in Urinary Excretion | Eight hours after first dose on Week 2 prior to first BCG instillation
  PK measurement expressed as cumulative fraction of dose in urinary excretion for APL-1202
Pharmacokinetics - Cumulative Fraction of Dose in Urinary Excretion | Eight hours after first dose on Week 6 prior to fifth BCG instillation
  PK measurement expressed as cumulative fraction of dose in urinary excretion for APL-1202

CONTACTS AND LOCATIONS:
Overall Officials: Harish Dave, MD, Study Chair — Linical Accelovance
Locations (2):
- United States (2):
  - The Icahn School of Medicine at Mt. Sinai, New York, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina

IPD SHARING:
Plan to Share IPD: No